CLINICAL TRIAL: NCT07060209
Title: A Randomized, Open-label, Single Oral Dose Clinical Trial to Evaluate the Food Effect on the Pharmacokinetics of Pelubiprofen-Tramadol (DW-1021) Controlled Release Film Coated Tablet (Pelubiprofen 45mg / Tramadol 45.9mg) After Oral Administration in 14 Healthy Adult Vietnamese Male Subjects Under Fed and Fasting Conditions
Brief Title: Food Effect on PK of DW-1021 (Pelubiprofen 45 mg / Tramadol 45.9 mg) in Healthy Adults
Acronym: DW-1021F
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Collaborators: Daewon Pharmaceutical Co., Ltd. (Industry); Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW-1021F; Protocol No. DW-1021F (Other: Daewon Pharmaceutical Co., Ltd.)
Record Dates: First submitted 2025-06-28; First posted 2025-07-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers; Pharmacokinetics; Food Effect in Healthy Volunteers
Keywords: Pelubiprofen; DW-1021; Tramadol; Food effect

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, two-period, two-sequence crossover design. Each subject will receive DW-1021 once under fasting conditions and once under fed conditions, with a 14-day washout period between periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DW-1021 Fasting Arm (Experimental): Subjects receive a single oral dose of DW-1021 under fasting conditions in Period 1 or Period 2 of the randomized two-period, two-sequence crossover design.
  Interventions: Drug: DW-1021
- DW-1021 Fed Arm (Experimental): Subjects receive a single oral dose of DW-1021 under fed conditions in Period 1 or Period 2 of the randomized two-period, two-sequence crossover design.
  Interventions: Drug: DW-1021

INTERVENTIONS:
Drug: DW-1021 — A fixed-dose combination controlled release film-coated tablet containing pelubiprofen 45 mg and tramadol 45.9 mg (salt form), administered as a single oral dose under fasting and fed conditions in a two-period, two-sequence crossover design. Each subject receives the intervention once under each condition with a 14-day washout period.

SUMMARY:
This is a Phase 1, open-label, single-dose crossover study designed to evaluate the effect of food on the pharmacokinetics of DW-1021, a fixed-dose combination tablet containing pelubiprofen 45 mg and tramadol 45.9 mg. Fourteen healthy adult Vietnamese males will each receive DW-1021 once under fasting conditions and once under fed conditions, with a 14-day washout period in between. Blood samples will be collected to assess how food intake affects the absorption and exposure levels of both active ingredients. Safety, including adverse events, laboratory results, vital signs, and ECGs, will be closely monitored throughout the study.

DETAILED DESCRIPTION:
DW-1021 is a fixed-dose combination tablet containing pelubiprofen, a nonsteroidal anti-inflammatory drug (NSAID), and tramadol, a centrally acting analgesic. Combining these two agents is expected to provide multimodal pain relief by targeting both peripheral and central pain pathways while potentially reducing opioid-related side effects.

This Phase 1 study is being conducted to evaluate how a standard high-fat meal affects the rate and extent of absorption of pelubiprofen and tramadol when administered together in DW-1021. A randomized, open-label, two-period, two-sequence crossover design is used to allow each subject to serve as his own control, improving the reliability of the pharmacokinetic comparison between fasting and fed states.

Each of the 14 healthy adult male volunteers will receive a single dose of DW-1021 under fasting conditions in one period and under fed conditions in the other, with a sufficient washout period to prevent carryover effects. Intensive blood sampling will be performed after each dose to measure plasma concentrations of pelubiprofen, its active metabolite (trans-OH-pelubiprofen), tramadol, and O-desmethyl-tramadol. Safety will be monitored throughout, including recording of adverse events, laboratory tests, vital signs, and ECGs.

The data generated will help determine whether food intake has a clinically significant impact on the pharmacokinetic profile of DW-1021 and will support future dosing recommendations and product labeling.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 20 to 40 years at screening visit
2. Body Mass Index (BMI) between 18.5 and 24.9 kg/m²
3. Body weight greater than 50 kg
4. Systolic blood pressure between 100 mmHg and 129 mmHg; diastolic blood pressure less than 84 mmHg
5. Regular heart rate ranging from 60 to 90 beats per minute
6. No clinically significant medical history or evidence of congenital or chronic diseases, including but not limited to: hypertension, orthostatic hypotension, hypoglycemia when fasting, swallowing difficulties, diabetes, cardiovascular diseases, pulmonary diseases, gastrointestinal diseases, liver insufficiency, renal insufficiency, endocrine disorders, neurological or psychiatric disorders, immunological, hematological, or hereditary diseases, tuberculosis, or infectious diseases
7. Suitable laboratory test results (hematology, urinalysis, blood chemistry, HCV/AIDS, HBsAg, anti-HCV) and electrocardiogram (ECG) at screening: no pathological findings; clinical laboratory parameters within the normal range or, if outside the normal range, not clinically significant as judged by the investigator
8. Willing and able to provide written informed consent after being fully informed about the study objectives and possible adverse effects
9. Agree to use effective contraception from initial administration until 7 days after the last dose of test or reference drugs

Exclusion Criteria:

1. Use of drugs that induce or inhibit drug-metabolizing enzymes (e.g., barbiturates) within 30 days prior to administration, or use of any medication that might affect the study within 10 days prior to administration
2. Participation in any other clinical trial within 3 months prior to screening
3. Blood donation within 8 weeks prior to drug administration
4. History of gastrointestinal surgery that may affect drug absorption
5. History of drug abuse, or use of alcohol, drugs, or tobacco products within 1 year before participation
6. Known hypersensitivity or allergy to the test or reference drug or their components
7. Known genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption, which are characterized by symptoms like diarrhea and bloating after consuming dairy products
8. Suffering from dysphagia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 48 hours post-dose in each period
  Cmax of pelubiprofen, tramadol will be assessed following a single oral administration of DW-1021 under fasting and fed conditions to evaluate the effect of food on systemic exposure.
Area Under the Concentration-Time Curve (AUC₀-t) | Up to 48 hours post-dose in each period
  AUC₀-t of pelubiprofen,tramadol will be assessed following a single oral administration of DW-1021 under fasting and fed conditions to evaluate the effect of food on systemic exposure.

SECONDARY OUTCOMES:
Cmax of trans-OH-pelubiprofen and O-desmethyl-tramadol | Up to 48 hours post-dose in each period
  Maximum observed plasma concentration (Cmax) of trans-OH-pelubiprofen and O-desmethyl-tramadol following single oral administration of DW-1021 under fasting or fed condition
AUC₀-t of trans-OH-pelubiprofen and O-desmethyl-tramadol | Up to 48 hours post-dose in each period
  Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC₀-t) for trans-OH-pelubiprofen and O-desmethyl-tramadol following single oral administration of DW-1021 under fasting or fed condition
Tmax of trans-OH-pelubiprofen and O-desmethyl-tramadol | Up to 48 hours post-dose in each period
  Time to reach maximum plasma concentration (Tmax) of trans-OH-pelubiprofen and O-desmethyl-tramadol following single oral administration of DW-1021 under fasting or fed condition.
t½ of trans-OH-pelubiprofen and O-desmethyl-tramadol | Up to 48 hours post-dose in each period
  Terminal elimination half-life (t½) of trans-OH-pelubiprofen and O-desmethyl-tramadol following single oral administration of DW-1021 under fasting or fed condition.
CL/F of trans-OH-pelubiprofen and O-desmethyl-tramadol | Up to 48 hours post-dose in each period
  Apparent oral clearance (CL/F) of trans-OH-pelubiprofen and O-desmethyl-tramadol following single oral administration of DW-1021 under fasting or fed condition

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial and Bioequivalence Center, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the limited scope of the Phase I pharmacokinetic study in healthy volunteers. The study does not include plans or infrastructure for external data sharing

REFERENCES:
- [Background] Shin JS, Baek SR, Sohn SI, Cho YW, Lee KT. Anti-inflammatory effect of pelubiprofen, 2-[4-(oxocyclohexylidenemethyl)-phenyl]propionic acid, mediated by dual suppression of COX activity and LPS-induced inflammatory gene expression via NF-kappaB inactivation. J Cell Biochem. 2011 Dec;112(12):3594-603. doi: 10.1002/jcb.23290. PMID 21809372
- [Background] Choi IA, Baek HJ, Cho CS, Lee YA, Chung WT, Park YE, Lee YJ, Park YB, Lee J, Lee SS, Yoo WH, Song JS, Kang SW, Kim HA, Song YW. Comparison of the efficacy and safety profiles of a pelubiprofen versus celecoxib in patients with rheumatoid arthritis: a 6-week, multicenter, randomized, double-blind, phase III, non-inferiority clinical trial. BMC Musculoskelet Disord. 2014 Nov 18;15:375. doi: 10.1186/1471-2474-15-375. PMID 25403311